CLINICAL TRIAL: NCT07053579
Title: Cross-cultural Adaptation and Validation of the Pediatric Chemotherapy-induced Neuropathy (P-CIN) for Chinese Pediatric Oncology Patients: A Multi-center Study
Brief Title: Cross-cultural Adaptation and Validation of the P-CIN for Chinese Pediatric Oncology Patients
Status: Completed | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Shanghai Children's Medical Center (Other); Shenzhen Children's Hospital (Other Government); The Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital (Unknown)
Responsible Party: Principal Investigator, Dr Eva Ho, Associate professor, The Hong Kong Polytechnic University
Other Study IDs: Validation study_P-CIN
Record Dates: First submitted 2025-06-18; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Cancer
Keywords: Chemotherapy induced peripheral neuropathy; Pediatric Chemotherapy-Induced Neuropathy; Pediatric oncology; Psychometrics; Validation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire: Participants completed the translated P-CIN, Wong-baker FACES Pain Rating scale for pain, and Chinese version of the Pediatric Quality of Life Inventory (PedsQL) Cancer Module for quality of life.

SUMMARY:
The goal of this study was to conduct a cross-cultural adaptation of the P-CIN into the Chinese context, assess its psychometric properties, and determine the cut-off value of CIPN among Chinese pediatric oncology patients.

Participants provided demographic and clinical characteristics, and complete the translated P-CIN, Wong-baker FACES Pain Rating scale for pain, and Chinese version of the Pediatric Quality of Life Inventory (PedsQL) Cancer Module for quality of life.

DETAILED DESCRIPTION:
A methodological, descriptive study was conducted.

ELIGIBILITY:
Inclusion Criteria:

* (1) 6 to 18 years of age
* (2) were diagnosed with cancer
* (3) had received or were currently receiving neurotoxic chemotherapy drugs (e.g., Vincristine, Cisplatin, Carboplatin, Oxaliplatin, Paclitaxel, Docetaxel, Ixabepilone, Bortezomib, Thalidomide)
* (4) were able to communicate, read, and write in Chinese without significant hearing and vision problems to ensure they understood the P-CIN.

Exclusion Criteria:

* (1) had a diagnosis of cancer in the central nervous system (CNS) cancer, cancer relapse or secondary cancer
* (2) in the terminal stage
* (3) planned to receive multiple cancer treatment (e.g., radiotherapy and immunotherapy)
* (4) suffered from other neuromuscular diseases (e.g., traumatic brain injury and cerebral palsy)
* (5) had a developmental deficit (e.g., Down's syndrome and other chromosomal disorders)
* (6) have suffered from psychiatric diseases or used antipsychotic drugs
* (7) had peripheral neuropathy symptoms caused by diabetes, genetic diseases, spinal cord injury, or alcoholism, or
* (8) had other neuromuscular disorders (e.g., traumatic brain injury, cerebral palsy).

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We recruited pediatric oncology patients from inpatient wards in Shenzhen Children's Hospital, Henan Cancer Hospital and Shanghai Children's Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Pediatric chemotherapy-induced peripheral neuropathy (P-CIN) scale | Baseline
  For measuring participants' peripheral neuropathy induced by chemotherapy. The total score ranges from 0 to 65 with higher scores indicating more severe chemotherpay induced peripheral neuropathy.

OTHER OUTCOMES:
Wong-baker Faces Pain Rating scale | Baseline
  For measuring participants' pain related to chemotherpay induced peripheral neuropathy.This scale contains six faces with increasing degree of pain from left to right, where each face is rated on a scale of 10, in which 0 indicates no hurt, 2 indicates little bit hurts, 4 indicates little more hurts, 6 indicates even more hurts, 8 indicated a whole lot of hurts, and 10 indicated the worst hurts. higher scores indicating more severe pain.
Chinese version of the Pediatric Quality of Life Inventory (PedsQL) Cancer Module | Baseline
  To assess the participants' quality of life. The participants rated how frequently a particular problem occurred in the past month, using a three-point Likert scale (0 = Not at all, 2 = Sometimes, 4 = A lot) for children 5-7 years old and a five-point Likert scale (0 = Never, 1=Almost never, 2=sometimes, 3=often, 4 = Almost always) for children of 8-18 years old and for the parents of patients of all ages. Each item score will be reversely scored and then linearly transformed into 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0). The scale score is the average of the total item scores, with higher scores representing better quality of life.
Clinician diagnosis of pediatric CIPN | Baseline
  To ascertain the clinical diagnosis of CIPN in participants. The clinical diagnosis of CIPN could be made if the results of the nerve conduction study are abnormal, with a score of the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) ≥ 2 after the clinical consultation with a pediatric neurologist on the chemotherapeutic drugs used, cumulative doses, and clinical characteristics and time course of the CIPN symptoms. NCI-CTCAE items including five items: peripheral sensory neuropathy, peripheral motor neuropathy, constipation, diarrhea, and neuralgia. The sum score for the five NCI-CTCAE items was between 0 and 17.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yan Ho, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - Ka Yan Ho, Hong Kong, China
  - The Hong Kong Polytechnic University, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT07053579/Prot_000.pdf
  • Informed Consent Form (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT07053579/ICF_001.pdf